CLINICAL TRIAL: NCT05397561
Title: Turkish Translation of Physical Activity Barriers and Facilitators Scale; Validity, Reliability, and Cultural Adaptation
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yunus Emre Tutuneken, Lecturer, Istinye University
Other Study IDs: 3
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Youth; Physical Activity; Physical Activity Barriers; Physical Activity Facilitators
Keywords: reliability; validity; facilitator; barrier; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Turkish Translation of Physical Activity Barriers and Facilitators Scale — Participants to be included in the study will be listed under a special code (traffic code of their city of birth, date of birth and order of participation). The socio-demographic characteristics, age, gender, body weight, height and Body Mass Index (BMI) of the participants will be evaluated and recorded with a specially prepared evaluation form. All participants in the study will complete the Turkish version of the PABFS, the Physical Activity Disability Scale (PADS), the Motivation for Participation in Physical Activity Scale (MPPAS), and the International Physical Activity Questionnaire (IPAQ) at their first visit. Participants will complete the BFYPA again after 7 days.

SUMMARY:
Background:The aim of our study is to examine the validity and reliability of the Turkish version of the "Barriers & Facilitators to Youth Physical Activity Questionnaire" in young individuals after cultural adaptation. The results of this study may shed light on youth PA participation studies, enable a clear explanation of the barriers and facilitators of physical activity in community-based research, and develop goal-oriented strategies for PA participation.

Material&Method: The research will be carried out at İstinye University and young individuals between the ages of 18-24, who accepted to participate in the study as a result of the invitation and whose family consent was obtained, will participate in the research. The socio-demographic characteristics, age, gender, body weight, height and Body Mass Index (BMI) of the participants will be evaluated and recorded with a specially prepared evaluation form. All participants in the study will complete the Turkish version of the BFYPA,The Exercise Benefits/Barriers Scale (EBBS), Motivation for Participation in Physical Activity Scale (MPPAS), and the International Physical Activity Questionnaire (IPAQ) at their first visit. Translation and cultural adaptation process of the original BFYPA Beaton et al. (2000) with reference to the guideline .

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18and 24
* Being Turkish literacy

Exclusion Criteria:

* Having neurological and musculoskeletal problems that can change physical activity habits, -Having heart and respiratory system problems,
* Having diabetes mellitus,
* Using chronic medication,
* Having a body mass index of 35 kg/m2 and being above,
* Any other condition that prevents physical activities.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy university students aged 18-24.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Physical Activity Barriers and Facilitators Scale (BFYPA) | 01.07.2022-01.07.2023
  Physical Activity Barriers and Facilitators Scale (Arlinghaus et al. 2021) consists of two subscales. Provides information on barriers and facilitators to physical activity among young people. BFFA is a Likert-type scale consisting of 20 items. Items were graded between 1-5 values corresponding to "Never" and "Always" . Written permission to use the scale was obtained for this study and the scale developers sent the scale.

SECONDARY OUTCOMES:
The Exercise Benefits/Barriers Scale (EBBS) | 01.07.2022-01.07.2023
  EBBS was developed to assess perceived benefits and perceived barriers to engaging in physical activity. The EBBS consists of two subscales and forty-three questions. Benefits are assessed by 29 items and barriers are assess by 14 items. Participants were asked to rate the perceived benefits and perceived barriers on a 4-point Likert Scale, with the response option ranging from "strongly agree= 4" to "strongly disagree = 1." The possible scores on the benefits scale ranged from 29 to 116 points, with higher scores indicating greater benefits. The possible range of scores on the barriers scale was 14 to 56 points, with a higher score indicating fewer perceived barriers.
Motivation Scale for Participation in Physical Activity (MSPPA) | 01.07.2022-01.07.2023
  Motivation Scale for Participation in Physical Activity was developed by Demir (2018) to measure high school students' motivation to participate in physical activity. MSPPA is a likert-type scale consisting of 16 items. The lowest score that can be obtained from the scale is 16, and the highest score is 80. The high scores of the participants on the scale mean that their motivation to participate in physical activity is positive. In this context, the scores obtained by the participants from the MSPPA indicate that they have 1-16 very low, 17-32 low, 33-48 medium, 49-64 high, 65-80 very high motivation to participate in physical activity. The Cronbach's alpha internal consistency coefficient of the original scale was found to be between 0.82 and 0.89. Spearman Brown split-half reliability coefficients were found to vary between 76 and 89.
Physical Activity Questionnaire (IPAQ) Short Form | 01.07.2022-01.07.2023
  The validity and reliability study of the International Physical Activity Questionnaire (IPAQ) in Turkey was carried out by Öztürk in 2005. In our study, the self-administered short form of the questionnaire with 7 questions covering the last 1 week will be used to evaluate the level of physical activity. Calculation of the total score of the short form includes the sum of time (minutes) and frequency (days) of walking, moderate-intensity activity, and vigorous activity. .

CONTACTS AND LOCATIONS:
Locations (1):
- Yunus Emre TÜTÜNEKEN, Istanbul, Zeytinburnu, Turkey (Türkiye)